CLINICAL TRIAL: NCT06009172
Title: The Effect of Auricular Point Acupressure on Sleep Quality in Women With Polycystic Ovary Syndrome：A Randomized Controlled Trial
Brief Title: APA on Sleep Quality in Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: XMYY-2022KY055-01
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA group (Experimental)
  Interventions: Other: Auricular point acupressure (APA)
- Control group (No Intervention)

INTERVENTIONS:
Other: Auricular point acupressure (APA) — Auricular point acupressure (APA) is a method derived from Traditional Chinese Medicine. PCOS women in the APA group began to apply pressure on the first day of enrollment. Patients were instructed to press each acupuncture point 3 times a day for 30 times. The PCOS woman is then trained to go to the outpatient clinic every 5-7 days to change the auricular acupressure sticker. The intervention period was 4 weeks.
  Arms: APA group

SUMMARY:
Women with polycystic ovary syndrome (PCOS) appear to have an increased frequency of sleep problems. The aim of this study was to explore the effect of auricular point acupressure (APA) pressure on sleep quality in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a prevalent disorder affecting 5-18% of reproductive-age women. In recent years, women with PCOS appear to have an increased frequency of sleep problems, and the prevalence of poor sleep in PCOS is high at 31%. The aim of this study was to explore the effect of auricular point acupressure (APA) pressure on sleep quality in women with PCOS. We verified the effect of APA pressure on sleep quality, quality of life, anxiety level, sex hormone indexes, and biochemical indexes in two groups after the intervention. So as to provide a sleep management strategy in PCOS women for future clinical practice guidelines.

ELIGIBILITY:
Subjects were included if they

1. were aged between 18-40 years old;
2. met the clinical diagnostic criteria of Western and Chinese medicine for PCOS with sleep disorders;
3. were evaluated by the Pittsburgh Sleep Quality Index Scale (PSQI) and had a score ≥ 7 points;
4. did not participate in other clinical trials.

Subjects were excluded if they

1. had a serious organic condition such as cardiovascular, cerebrovascular, liver, or kidney disease;
2. had acute gynecological inflammation, gynecological tumors, or reproductive system malformations;
3. had severe anxiety, depression, or other mental illnesses;
4. were pregnant;
5. had used sleeping and sedative drugs in the past month;
6. were allergic to ear point tape;
7. had local rupture of the skin at the selected ear point;
8. refused to fill out questionnaires and sign informed consent forms.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 30 days
  The PSQI is a cornerstone tool for the assessment of sleep quality

SECONDARY OUTCOMES:
Modified Polycystic Ovary Syndrome Health Related Quality of Life Questionnaire (MPCOSQ) | Baseline and 30 days
Self-Rating Anxiety Scale (SAS) | Baseline and 30 days
  The cutoff value for anxiety assessment of Self-Rating Anxiety Scale (SAS) is 50 oints, and the higher the score, the more obvious the anxiety tendency. Below 49 is normal; 50-59 is mild; 60-69 is moderate; A score of 69 or above is considered severe.
Testosterone (T) level(ng/mL） | Baseline and 30 days
Progesterone (P) level(ng/mL） | Baseline and 30 days
fasting serum insulin (pmol/L) | Baseline and 30 days
fasting blood-glucose(mmol/L) | Baseline and 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Diabetes, the First Affiliated Hospital of Xiamen University, School of medicine, Xiamen university, Xiamen, China, Xiamen, Fujian, China